CLINICAL TRIAL: NCT05034575
Title: A Study to Assess Eye Tracking and Visual Gaze Patterns in Laryngology
Brief Title: Eye Tracking in Laryngology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diana M. Orbelo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-012365
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novice and experienced medical personnel (Experimental): Participants will be asked to complete two tasks each taking approximately 10 minutes while wearing eye-tracking technology to understand focus of gaze during laryngeal endoscopy and stroboscopy interpretation.
  Interventions: Other: Eye Tracking Technology Sensor

INTERVENTIONS:
Other: Eye Tracking Technology Sensor — Eye tracking will be performed using Tobii Pro eye tracking technology sensor (Tobii Pro Fusion, Stockholm, Sweden), providing binocular eye tracking up to 250 Hz. The sensor, positioned on the inferior aspect of the computer monitor, reflects infrared (IR) light beams off of each cornea and are subsequently captured.

SUMMARY:
The purpose of this study is to assess whether eye-tracking technology can be used to differentiate the visual gaze patterns of experienced and novice laryngoscopists while reviewing prerecorded laryngeal videos with both normal and abnormal findings and to characterize any differences arising between level of training groups.

DETAILED DESCRIPTION:
Novice and experienced participants will be recruited to take part in this study. Novices include medical students without practical experience in otorhinolaryngology and resident physicians at different stages in training. Trainees, residents and experts from fields of gastroenterology and pulmonology will also be included. The experienced group will be defined as consultants and speech pathologists.

This study will look at multiple areas within otolaryngology including laryngology, rhinology, facial plastic surgery, head and neck oncology, and otology. Participants will view prerecorded videos and/or still pictures absent of patient identifiers.

There will be two tasks each taking approximately 10 minutes. Task order will be alternated between subjects with one task asking participants to view 7 still images from video laryngoscopy examinations. After each image participants will rate how likely the image is to represent glottic cancer and what portion of the image they deemed most important to their decision. For the second task, participants will be asked to view a 5 second video of a flexible laryngoscope exam, after which, they will be asked to identify the presence and side of vocal fold paralysis as well as note the location they deemed most important to their decision.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and over.
* Already professionals in a laryngology related field, residents in a related field or students considering a related field.
* Related fields include otolaryngology, laryngology, and speech language pathology.

Exclusion Criteria:

- Anyone not meeting the inclusion criteria or anyone not wishing to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Time to Fixation Fixation Point | 15 minutes
  Defined as the temporary suspension of eye movement (80ms) on a specific point (≤ 30 pixels) within the field of view.
Percent of Fixation Time on pre determined area of interest | 15 minutes
  Defined as the percent of total gaze time on area of interest
Count of Fixations | 15 minutes
  Number of times observer returns gaze to area of interest

CONTACTS AND LOCATIONS:
Overall Officials: Diana Orbelo, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials